CLINICAL TRIAL: NCT01351896
Title: Phase II Study of Lenalidomide to Repair Immune Synapse Response and Humoral Immunity in Early-Stage, Asymptomatic Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) With High-Risk Genomic Features
Brief Title: Lenalidomide and Vaccine Therapy in Treating Patients With Early-Stage Asymptomatic Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02584; NCI-2011-02584 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000698438; OSU 10156; 2011C0005; 8834 (Other: Ohio State University Comprehensive Cancer Center); 8834 (Other: CTEP); N01CM00070 (NIH); N01CM62207 (NIH); P01CA095426 (NIH); P30CA016058 (NIH); P50CA140158 (NIH)
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Results first posted 2025-08-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Ann Arbor Stage I Small Lymphocytic Lymphoma; Ann Arbor Stage II Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia With Unmutated Immunoglobulin Heavy Chain Variable-Region Gene; Small Lymphocytic Lymphoma; Small Lymphocytic Lymphoma With Unmutated Immunoglobulin Heavy Chain Variable-Region Gene; Stage 0 Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Specimen Handling; Biopsy; Lenalidomide; Pneumococcal Vaccines; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Concurrent PCV13 and lenalidomide) (Experimental): Patients receive low-dose lenalidomide PO once daily on days 1-28. Treatment repeats every 28 days for at least 24 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive PCV13 IM on day 1 of courses 3 and 5.
  Patients may undergo bone marrow biopsy and aspirate and CT during screening and blood sample collection throughout the study. (Blood sample collection discontinued with approval of protocol version 24 dated 3/15/2024)
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Lenalidomide; Biological: Pneumococcal Polyvalent Vaccine
- Arm B (Sequential PCV13 and lenalidomide) (Experimental): Patients receive PCV13 IM on days 1 and 78 (cycles 1 and 3). Patients also receive low-dose lenalidomide as in arm 1 beginning on day 1 of course 4. Treatment repeats every 28 days for at least 24 cycles in the absence of disease progression or unacceptable toxicity. Patients may undergo bone marrow biopsy and aspirate and CT during screening and blood sample collection throughout the study. (Blood sample collection discontinued with approval of protocol version 24 dated 3/15/2024)
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Lenalidomide; Biological: Pneumococcal Polyvalent Vaccine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Biological: Pneumococcal Polyvalent Vaccine — Given IM (concurrently or sequentially)
  Other Names: PCV 23; Pneumococcal 23-valent Polysaccharide Vaccine; Pneumococcal Polysaccharide Vaccine; Pneumococcal Vaccine Polyvalent; Pneumovax 23; Pnu-Imune 23; PPSV; PPSV23; PPSV23 Vaccine

SUMMARY:
This phase II trial studies the effect of lenalidomide and vaccine in treating patients with early-stage asymptomatic chronic lymphocytic leukemia or small lymphocytic lymphoma. Lenalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. It may also stimulate the immune system in different ways and stop cancer cells from growing. Vaccines may help the body build an effective immune response to kill cancer cells. Giving lenalidomide together with vaccine therapy may make a stronger immune response and kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the proportion of early-stage, high-risk chronic lymphocytic leukemia (CLL) patients achieving a response (>= 4-fold increase from baseline and/or antibody concentrations >= 0.35 ug/mL in 6 of 7 type-specific anti-pneumococcal antibody levels) after 2 doses of pneumococcal 13-valent conjugated vaccine (Prevnar 13, PCV13 [pneumococcal polyvalent vaccine]) administered concurrent with versus sequential to low-dose lenalidomide.

SECONDARY OBJECTIVES:

I. To determine the complete response (CR) rate after 2 years of lenalidomide therapy.

II. To determine the time to first treatment (TFT), defined as the time from diagnosis to first non-lenalidomide therapy for progressive CLL as described by International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria.

III. To determine the incidence of infection and invasive pneumococcal infections following treatment with the PCV13 vaccine and either concurrent or sequential lenalidomide.

IV. To determine the frequency of humoral and cellular immune response to CLL tumor antigens following treatment with the PCV13 vaccine and either concurrent or sequential lenalidomide.

V. To determine the safety and toxicity associated with long-term lenalidomide exposure.

VI. To perform correlative pharmacodynamic and pharmacokinetic studies and correlate these with vaccine/tumor immunologic and disease response.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A (concurrent PCV13 and lenalidomide): Patients receive low-dose lenalidomide orally (PO) once daily on days 1-28. Treatment repeats every 28 days for at least 24 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive 13-valent protein-conjugated pneumococcal vaccine (PCV13) intramuscularly (IM) on day 1 of courses 3 and 5.

ARM B (sequential PCV13 and lenalidomide): Patients receive PCV13 IM on days 1 and 78 (cycles 1 and 3). Patients also receive low-dose lenalidomide as in arm 1 beginning on day 1 of cycle 4. Treatment repeats every 28 days for at least 24 cycles in the absence of disease progression or unacceptable toxicity.

Patients may undergo bone marrow biopsy and aspirate and computed tomography (CT) during screening and blood sample collection throughout the study. (Blood sample collection discontinued with approval of protocol version 24 dated 3/15/2024)

After completion of study treatment, patients are followed up for 30 days, every 3 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically identified chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) as defined by the World Health Organization (WHO) classification of hematopoietic neoplasms
* CLL/SLL cells must demonstrate one or more of the following high-risk genomic features:

  * Deletion (Del) (17p13.1) as detected by fluorescence in-situ hybridization (FISH) in > 20% of cells
  * Del(11q22.3) as detected by FISH in > 20% of cells
  * Complex karyotype (>= 3 cytogenetic abnormalities on stimulated karyotype)
  * Unmutated immunoglobulin variable heavy chain (IgVH) (>= 98% sequence homology compared with germline sequence)
* Patients cannot meet any of the following consensus criteria for initiating treatment:

  * Progressive splenomegaly and/or lymphadenopathy identified by physical examination or radiographic studies
  * Progressive lymphocytosis with total white blood cell (WBC) >= 300,000/uL
  * Anemia (< 11 g/dL) or thrombocytopenia (< 100,000/uL) due to bone marrow involvement
  * Presence of unintentional weight loss > 10% over the preceding 6 months
  * National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or 3 fatigue
  * Fevers > 100.5 degrees or night sweats for > 2 weeks without evidence of infection
  * Progressive lymphocytosis with an increase of > 50% over a 2 month period or an anticipated doubling time of < 6 months
* No prior therapy for CLL/SLL, including chemotherapy, radiotherapy, and/or immunotherapy will be allowed
* Age ≥ 18 years and < 80 years (or with justification if older than 80 years due to the higher risk of toxicity in patients older than 80 years). CLL is rare in children and likely represents a different disease process. As a result, children are excluded from this study but may be eligible for future pediatric phase 2 combination trials
* Estimated life expectancy of greater than 24 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Total bilirubin =< 1.5 times upper limit of normal (ULN) (unless secondary to Gilbert disease)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate-pyruvate transaminase [SGPT]) =< 2.5 times ULN
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal according to the Cockcroft-Gault formula
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelet count >= 100,000/uL
* Able to swallow capsules without difficulty and no history of malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide. Further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure

Exclusion Criteria:

* Patients who have had any treatment for their CLL/SLL, including but not limited to chemotherapy, radiotherapy, or immunotherapy, prior to entering the study
* No corticosteroid use will be permitted within two weeks prior to study, except for maintenance therapy for a non-malignant disease; maintenance therapy dose may not exceed 20 mg/day prednisone or equivalent
* Patients who meet consensus criteria for the treatment of CLL/SLL
* Patients may not be receiving any other investigational agents
* Patients with a recent history (within 6 months of study entry) of deep vein thrombosis (DVT)/pulmonary embolism (PE) are not eligible; patients with a distant history (greater than 6 months before study entry) of venous thromboembolic disease are eligible, but should receive prophylactic aspirin or low molecular weight heparin
* History of allergic reactions attributable to compounds of similar chemical or biologic composition to thalidomide, lenalidomide or any component of PCV7 or PCV13, including the diphtheria toxoid
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject is considered by his or her physician to have a 2 year survival expectation
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because lenalidomide is an immunomodulatory agent (IMID) with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide, breastfeeding should be discontinued if the mother is treated with lenalidomide
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy will be eligible if they otherwise meet required hematologic parameters and are not receiving an antiviral agent with known or potential interaction with lenalidomide; because the primary aim of this study is to measure the immune response to pneumococcal vaccination, only patients with CD4 cell counts >= 200 and viral load < 50 will be eligible
* Patients who have been treated for autoimmune hemolytic anemia or autoimmune thrombocytopenia within the last 6 months or are direct antiglobulin test/Coombs test or indirect antiglobulin test positive at the time of screening
* Patients who have developed erythema nodosum characterized by a desquamating rash while taking thalidomide or similar drugs in the past are excluded
* Because of the potential for H2-blockers to modulate antibody response to pneumococcal vaccine, patients must discontinue treatment with H2-blockers (cimetidine, ranitidine, etc.) prior to beginning protocol therapy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-11-02 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2026-05-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Rogers, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Concurrent PCV13 and Lenalidomide): Patients receive low-dose lenalidomide PO once daily on days 1-28. Treatment repeats every 28 days for at least 24 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive PCV13 IM on day 1 of courses 3 and 5.
  Patients may undergo bone marrow biopsy and aspirate and CT during screening and blood sample collection throughout the study. (Blood sample collection discontinued with approval of protocol version 24 dated 3/15/2024)
  Biospecimen Collection: Undergo blood sample collection
  Bone Marrow Aspiration: Undergo bone marrow aspiration
  Bone Marrow Biopsy: Undergo bone marrow biopsy
  Computed Tomography: Undergo CT
  Lenalidomide: Given PO
  Pneumococcal Polyvalent Vaccine: Given IM (concurrently or sequentially)
Period: Overall Study
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Started | 24 | 25
Completed | 24 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide) | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Median (Full Range); unit: years] | 61 [48 to 69] | 57 [40 to 70] | 59 [40 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 16 | 18 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 22 | 25 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Achieve an Antibody Response
Description: Defined as achieving at least a four-fold increase in post-vaccination serotype-specific immunoglobulin G (IgG) titers or serotype-specific IgG concentrations of >= 0.35 ug/mL for 6 of 7 serotypes measured by a standard enzyme linked immunosorbent assay.
Time Frame: Up to 1 month
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
percentage of participants | 75 | 88

2. Secondary Outcome: Seroconversion Rates
Description: Summarized using descriptive statistics by treatment arm.
Time Frame: Up to 4 years
Reporting Status: Not Posted

3. Secondary Outcome: Complete Response Rate
Description: 95% confidence intervals will be estimated. A designation of complete response (CR) requires all of the following for a period of at least two months from completion of therapy:
  * Absence of adenopathy on physical exam.
  * No hepatomegaly or splenomegaly on physical exam.
  * Absence of constitutional symptoms.
  * Normal CBC as exhibited by polymorphonuclear leukocytes ≥ 1500/µL, platelets > 100,000/µL, hemoglobin > 11.0 g/dL (untransfused), and lymphocyte count < 5,000/ µL.
  * Bone marrow aspirate and biopsy must be normocellular for age with < 30% of nucleated cells being lymphocytes. Lymphoid nodules must be absent. If the marrow is hypocellular, a repeat determination should be performed in one month.
Time Frame: At 2 years
Population: The number of participants analyzed for complete response at 2 years is the number of participants for whom response data was available at the 2 year mark.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 16 | 20
percentage of participants | 6 [0.2 to 30] | 0 [0 to 17]

4. Secondary Outcome: Time to First Treatment
Description: Defined by International Workshop on chronic lymphocytic leukemia (CLL) (IWCLL) 2008 criteria. Summarized and explored between treatment arms using Kaplan-Meier methods. Reported as the probability of not starting the next treatment and its 95% CI for each year.
Time Frame: From study entry to first therapy for progressive CLL, assessed up to 4 years
Measure: Number (95% Confidence Interval); unit: probabibility rate
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
probabibility rate
  Year 1 | 0.88 [0.66 to 0.96] | 0.96 [0.75 to 0.99]
  Year 2 | 0.79 [0.57 to 0.91] | 0.92 [0.72 to 0.98]
  Year 3 | 0.79 [0.57 to 0.91] | 0.80 [0.58 to 0.91]
  Year 4 | 0.74 [0.51 to 0.88] | 0.70 [0.46 to 0.85]

5. Secondary Outcome: Overall Survival
Description: Summarized and explored between treatment arms using Kaplan-Meier methods.
Time Frame: Up to 4 years
Reporting Status: Not Posted

6. Secondary Outcome: Progression-free Survival
Description: Defined by International Workshop on chronic lymphocytic leukemia (CLL) (IWCLL) 2008 criteria. Summarized and explored between treatment arms using Kaplan-Meier methods.
Time Frame: Time from start of treatment to time of disease progression or death secondary to any cause, assessed up to 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Number of Adverse Events
Description: Summarized by and across treatment arms, along with the type, severity, and perceived attribution to study according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5. The rates of severe (grade 3+) toxicity (at least possibly related to treatment) and non-hematologic toxicity will be summarized; assuming the incidence of severe toxicity is binomially distributed, 95% confidence intervals will be calculated. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine the toxicity patterns. Adverse events occurring in greater than 5% of the participants in each arm will be reported in this outcome measure.
Time Frame: Up to 4 years
Measure: Number; unit: Number of Events
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
Number of Events
  Anemia | 46 | 38
  Leukocytosis | 3 | 9
  Lymph node pain | 7 | 10
  Cardiac disorders, other | 2 | 2
  Palpitations | 0 | 3
  Sinus bradycardia | 18 | 21
  Sinus tachycardia | 2 | 2
  Ear and labyrinth disorders, other | 1 | 3
  Ear pain | 1 | 4
  Tinnitus | 1 | 2
  Vertigo | 1 | 2
  Dry eye | 2 | 1
  Eye disorders, other | 1 | 4
  Floaters | 2 | 1
  Abdominal pain | 3 | 12
  Bloating | 1 | 7
  Constipation | 14 | 16
  Dental caries | 0 | 4
  Diarrhea | 42 | 63
  Dyspepsia | 2 | 7
  Flatulence | 3 | 1
  Gastroesophageal reflux disease | 5 | 3
  Gastrointestinal disorders, other | 4 | 5
  Mucositis oral | 0 | 6
  Nausea | 10 | 16
  Oral pain | 4 | 5
  Toothache | 2 | 2
  Vomiting | 2 | 8
  Chills | 2 | 0
  Edema limbs | 3 | 4
  Fatigue | 11 | 21
  Fever | 6 | 9
  Flu like symptoms | 4 | 2
  Localized edema | 7 | 9
  Non-cardiac chest pain | 3 | 3
  Pain | 9 | 8
  Gallbladder pain | 3 | 0
  Bronchial infection | 1 | 4
  Infections and infestations, other | 4 | 5
  Lung infection | 9 | 1
  Nail infection | 2 | 3
  Papulopustular rash | 1 | 2
  Prostate infection | 0 | 2
  Sinusitis | 10 | 9
  Skin infection | 7 | 2
  Upper respiratory infection | 23 | 21
  Urinary tract infection | 5 | 4
  Vaginal infection | 3 | 0
  Bruising | 4 | 14
  Fall | 3 | 8
  Injury, poisoning and procedural complications, other | 2 | 0
  Alanine aminotransferase increased | 28 | 34
  Alkaline phosphatase increased | 10 | 7
  Aspartate aminotransferase increased | 28 | 27
  Blood bilirubin increased | 25 | 37
  Creatinine increased | 29 | 26
  Hemoglobin increased | 0 | 3
  Lymphocyte count decreased | 25 | 21
  Lymphocyte count increased | 25 | 35
  Neutrophil count decreased | 119 | 100
  Platelet count decreased | 67 | 66
  Weight gain | 2 | 2
  Weight loss | 7 | 13
  White blood cell decreased | 57 | 28
  Anorexia | 1 | 3
  Dehydration | 4 | 1
  Hypercalcemia | 4 | 7
  Hyperglycemia | 94 | 117
  Hyperkalemia | 2 | 6
  Hypernatremia | 1 | 2
  Hyperuricemia | 14 | 37
  Hypoalbuminemia | 3 | 12
  Hypocalcemia | 22 | 18
  Hypoglycemia | 7 | 18
  Hypokalemia | 28 | 22
  Hypomagnesemia | 2 | 3
  Hyponatremia | 8 | 11
  Hypophosphatemia | 15 | 58
  Metabolism and nutrition disorders, other | 0 | 2
  Arthralgia | 7 | 10
  Arthritis | 1 | 2
  Back pain | 10 | 7
  Musculoskeletal and connective tissue disorder, other | 4 | 3
  Myalgia | 9 | 14
  Pain in extremity | 4 | 8
  Neoplasms, benign, malignant and unspecified, other | 6 | 10
  Dizziness | 7 | 10
  Dysesthesia | 11 | 9
  Dysgeusia | 3 | 1
  Headache | 19 | 29
  Paresthesia | 5 | 5
  Presyncope | 3 | 3
  Sinus pain | 0 | 2
  Anxiety | 0 | 2
  Confusion | 2 | 2
  Depression | 0 | 2
  Insomnia | 5 | 5
  Chronic kidney disease | 6 | 2
  Hematuria | 0 | 2
  Renal calculi | 0 | 2
  Allergic rhinitis | 13 | 10
  Cough | 14 | 27
  Dyspnea | 9 | 15
  Epistaxis | 2 | 1
  Hoarseness | 1 | 3
  Laryngeal inflammation | 1 | 2
  Nasal congestion | 7 | 5
  Postnasal drip | 1 | 12
  Productive cough | 6 | 10
  Respiratory, thoracic and mediastinal disorders, other | 1 | 6
  Sore throat | 11 | 20
  Hyperhidrosis | 1 | 5
  Pruritus | 3 | 2
  Rash acneiform | 6 | 0
  Rash maculo-papular | 27 | 19
  Skin and subcutaneous tissue disorders, other | 40 | 32
  Flushing | 2 | 2
  Hypertension | 80 | 90

8. Secondary Outcome: Pharmacokinetic (PK) Parameters of Lenalidomide
Description: PK will be graphically evaluated within and across arms to assess potential patterns and relationships.
Time Frame: Baseline, days 1 and 2 of course 2 (Arm A) and days 1 and 2 of course 5 (Arm B)
Reporting Status: Not Posted

9. Secondary Outcome: Change in Serum Immunoglobulin
Description: Pharmacodynamic markers will be graphically evaluated within and across arms to assess potential patterns and relationships.
Time Frame: Baseline up to 4 years
Reporting Status: Not Posted

10. Secondary Outcome: Change in Anti-tumor Antibody Levels
Description: as for outcome 9
Time Frame: Baseline up to 4 years
Reporting Status: Not Posted

11. Secondary Outcome: Antibody Titre Levels for Serotype 1
Description: Summarized using descriptive statistics by treatment arm. Changes in serotype-specific markers will be graphically evaluated between the two arms and the nonparametric Mann-Whitney rank sum test will be used to compare the geometric mean concentrations.
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: Participants in arm A were analyzed on cycle 1 day 1 (c1d1), c3d1, c5d1, and c6d1. Participants in arm B were analyzed on c1d1, c3d1, c4d1, and c10d1.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 4.1 (8.1) | 7.4 (15.2)
  Cycle 3 day 1 | 13.8 (47.1) | 10.1 (18.7)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 17.2 (28.2)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 18.2 (56.1) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 16.9 (45.0) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 7.9 (10.4)

12. Secondary Outcome: Antibody Titre Levels for Serotype 2
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 1.8 (2.0) | 1.5 (1.2)
  Cycle 3 day 1 | 1.7 (2.0) | 1.7 (1.8)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 1.8 (1.7)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 2.5 (3.0) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 2.0 (2.3) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 1.6 (1.2)

13. Secondary Outcome: Antibody Titre Levels for Serotype 3
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 2.0 (1.6) | 2.9 (5.4)
  Cycle 3 day 1 | 2.1 (2.0) | 11.1 (32.0)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 20.1 (58.0)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 3.0 (2.6) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 9.5 (12.3) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 6.5 (14.6)

14. Secondary Outcome: Antibody Titre Levels for Serotype 4
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 0.5 (0.5) | 1.4 (2.0)
  Cycle 3 day 1 | 0.6 (0.6) | 11.8 (50.8)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 18.3 (53.1)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 0.9 (0.9) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 6.1 (11.8) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 8.9 (25.1)

15. Secondary Outcome: Antibody Titre Levels for Serotype 5
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 2.7 (2.6) | 4.4 (5.8)
  Cycle 3 day 1 | 3.0 (2.8) | 16.0 (26.4)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 27.0 (39.6)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 11.0 (23.3) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 12.9 (17.2) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 30.1 (52.8)

16. Secondary Outcome: Antibody Titre Levels for Serotype 8
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 2.3 (3.0) | 2.0 (2.0)
  Cycle 3 day 1 | 2.1 (2.5) | 3.2 (5.5)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 3.4 (6.6)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 2.9 (3.7) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 2.2 (2.5) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 2.1 (2.4)

17. Secondary Outcome: Antibody Titre Levels for Serotype 9N
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 1.7 (1.5) | 2.9 (3.5)
  Cycle 3 day 1 | 2.0 (2.4) | 5.2 (12.5)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 8.7 (24.5)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 2.7 (3.9) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 3.1 (4.9) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 5.3 (10.8)

18. Secondary Outcome: Antibody Titre Levels for Serotype 12F
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 0.7 (0.8) | 0.9 (1.1)
  Cycle 3 day 1 | 0.7 (0.8) | 1.3 (1.4)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 1.2 (1.4)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 0.9 (0.9) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 0.7 (0.6) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 0.9 (0.9)

19. Secondary Outcome: Antibody Titre Levels for Serotype 14
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 0.5 (0.5) | 1.4 (2.0)
  Cycle 3 day 1 | 0.6 (0.6) | 11.8 (50.8)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 18.3 (53.1)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 0.9 (0.9) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 6.1 (11.8) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 8.9 (25.1)

20. Secondary Outcome: Antibody Titre Levels for Serotype 17F
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 9.7 (15.1) | 5.2 (5.7)
  Cycle 3 day 1 | 9.0 (13.2) | 6.0 (8.7)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 6.0 (8.5)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 14.4 (20.2) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 11.6 (18.4) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 4.2 (5.0)

21. Secondary Outcome: Antibody Titre Levels for Serotype 19F
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 3.5 (3.6) | 6.1 (15.3)
  Cycle 3 day 1 | 6.3 (14.2) | 13.3 (29.6)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 34.5 (68.8)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 13.6 (24.1) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 24.7 (37.0) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 14.7 (20.3)

22. Secondary Outcome: Antibody Titre Levels for Serotype 20
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 2.0 (4.4) | 1.9 (2.3)
  Cycle 3 day 1 | 1.9 (3.9) | 1.8 (2.2)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 2.1 (2.1)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 3.2 (5.5) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 2.1 (3.8) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 1.5 (1.6)

23. Secondary Outcome: Antibody Titre Levels for Serotype 22F
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 8.0 (7.7) | 10.2 (11.8)
  Cycle 3 day 1 | 9.2 (12.9) | 11.1 (16.7)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 11.5 (16.0)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 11.9 (16.8) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 10.7 (15.3) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 10.3 (14.8)

24. Secondary Outcome: Antibody Titre Levels for Serotype 23F
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 10.2 (14.6) | 15.9 (26.7)
  Cycle 3 day 1 | 9.4 (12.1) | 31.5 (51.2)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 45.3 (76.2)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 12.7 (17.2) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 17.0 (24.8) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 23.8 (38.9)

25. Secondary Outcome: Antibody Titre Levels for Serotype 6B
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 3.0 (2.9) | 6.7 (9.1)
  Cycle 3 day 1 | 4.2 (5.0) | 38.8 (101.9)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 60.2 (114.4)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 9.0 (14.4) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 17.8 (26.5) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 31.9 (50.6)

26. Secondary Outcome: Antibody Titre Levels for Serotype 10A
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 5.5 (11.6) | 4.7 (5.7)
  Cycle 3 day 1 | 6.7 (14.2) | 5.0 (5.7)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 4.7 (5.4)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 8.6 (15.5) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 6.9 (12.9) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 4.2 (5.1)

27. Secondary Outcome: Antibody Titre Levels for Serotype 11A
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 2.1 (2.8) | 1.5 (1.6)
  Cycle 3 day 1 | 2.0 (2.7) | 1.6 (1.7)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 1.8 (2.0)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 2.3 (2.9) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 1.9 (2.2) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 1.7 (2.3)

28. Secondary Outcome: Antibody Titre Levels for Serotype 7F
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 5.1 (6.6) | 7.6 (15.7)
  Cycle 3 day 1 | 4.9 (6.3) | 9.9 (20.1)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 17.0 (47.1)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 6.4 (6.0) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 5.7 (5.3) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 12.2 (25.8)

29. Secondary Outcome: Antibody Titre Levels for Serotype 15B
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 3.2 (6.9) | 4.4 (12.9)
  Cycle 3 day 1 | 3.3 (8.1) | 4.0 (10.2)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 4.7 (13.1)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 4.3 (8.2) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 3.7 (6.7) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 4.2 (11.0)

30. Secondary Outcome: Antibody Titre Levels for Serotype 18C
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 2.6 (4.8) | 3.8 (7.9)
  Cycle 3 day 1 | 3.8 (9.6) | 5.6 (8.8)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 10.6 (21.1)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 3.5 (4.9) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 9.6 (25.6) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 6.7 (14.6)

31. Secondary Outcome: Antibody Titre Levels for Serotype 19A
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 6.9 (10.4) | 7.0 (10.6)
  Cycle 3 day 1 | 5.3 (7.4) | 21.7 (63.4)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 37.0 (92.9)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 9.2 (9.6) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 12.2 (13.6) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 18.8 (35.7)

32. Secondary Outcome: Antibody Titre Levels for Serotype 9V
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 3.7 (5.6) | 4.5 (5.4)
  Cycle 3 day 1 | 4.0 (7.0) | 13.5 (30.1)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 14.1 (32.8)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 7.0 (13.3) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 6.3 (11.0) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 15.5 (28.2)

33. Secondary Outcome: Antibody Titre Levels for Serotype 33F
Description: as for outcome 11
Time Frame: Up to cycle 10 day 1 (each cycle is 28 days)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
Number analyzed (Participants) | 24 | 25
micrograms per milliliter
  Cycle 1 day 1 | 2.1 (2.6) | 2.2 (2.7)
  Cycle 3 day 1 | 2.1 (2.6) | 2.6 (3.6)
  Cycle 4 day 1: number analyzed (Participants) | 0 | 25
  Cycle 4 day 1 |  | 2.7 (3.8)
  Cycle 5 day 1: number analyzed (Participants) | 24 | 0
  Cycle 5 day 1 | 2.7 (3.2) |
  Cycle 6 day 1: number analyzed (Participants) | 24 | 0
  Cycle 6 day 1 | 2.1 (2.2) |
  Cycle 10 day 1: number analyzed (Participants) | 0 | 25
  Cycle 10 day 1 |  | 2.3 (3.2)

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Arm A (Concurrent PCV13 and Lenalidomide) | Arm B (Sequential PCV13 and Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 0/24 | 1/25
Serious Adverse Events (participants affected / at risk) | 12/24 | 13/25
Other Adverse Events (participants affected / at risk) | 24/24 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Concurrent PCV13 and Lenalidomide) (N=24) | Arm B (Sequential PCV13 and Lenalidomide) (N=25)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (3)
Chest pain- cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 3 (3) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase increased (Investigations) | 0 (0) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Creatinine Increased (Investigations) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified, other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Concurrent PCV13 and Lenalidomide) (N=24) | Arm B (Sequential PCV13 and Lenalidomide) (N=25)
Anemia (Blood and lymphatic system disorders) | 14 (46) | 15 (38)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3) | 5 (9)
Lymph node pain (Blood and lymphatic system disorders) | 6 (7) | 8 (10)
Cardiac disorders- other (Cardiac disorders) | 2 (2) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 9 (18) | 7 (21)
Sinus Tachycardia (Cardiac disorders) | 2 (2) | 1 (2)
Ear and labyrinth disorders, other (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Eye disorders, other (Eye disorders) | 1 (1) | 4 (4)
Floaters (Eye disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 6 (10)
Bloating (Gastrointestinal disorders) | 1 (1) | 4 (7)
Constipation (Gastrointestinal disorders) | 6 (14) | 11 (16)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 17 (41) | 21 (63)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (7)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (5) | 2 (3)
Gastrointestinal disorders, other (Gastrointestinal disorders) | 4 (4) | 3 (5)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 5 (6)
Nausea (Gastrointestinal disorders) | 5 (10) | 9 (16)
Oral pain (Gastrointestinal disorders) | 3 (4) | 5 (5)
Toothache (Gastrointestinal disorders) | 1 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (8)
Chills (General disorders) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 3 (3) | 3 (4)
Fatigue (General disorders) | 10 (11) | 19 (21)
Fever (General disorders) | 5 (5) | 7 (7)
Flu like symptoms (General disorders) | 4 (4) | 2 (2)
Localized edema (General disorders) | 6 (7) | 5 (9)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (3)
Pain (General disorders) | 9 (9) | 7 (8)
Gallbladder pain (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 3 (4)
Infections and infestations, other (Infections and infestations) | 3 (4) | 5 (5)
Lung infection (Infections and infestations) | 6 (6) | 1 (1)
Nail infection (Infections and infestations) | 2 (2) | 2 (3)
Papulopustular rash (Infections and infestations) | 1 (1) | 2 (2)
Prostate infection (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 6 (10) | 5 (9)
Skin infection (Infections and infestations) | 6 (7) | 2 (2)
Upper respiratory infection (Infections and infestations) | 13 (23) | 15 (21)
Urinary tract infection (Infections and infestations) | 3 (4) | 3 (4)
Vaginal infection (Infections and infestations) | 2 (3) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 4 (4) | 9 (14)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 7 (8)
Injury, poisoning and procedural complications, other (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 10 (28) | 15 (31)
Alkaline Phosphatase Increased (Investigations) | 4 (10) | 5 (7)
Aspartate Aminotransferase Increased (Investigations) | 10 (28) | 13 (24)
Blood bilirubin increased (Investigations) | 5 (25) | 7 (37)
Creatinine increased (Investigations) | 8 (28) | 5 (26)
Hemoglobin increased (Investigations) | 0 (0) | 2 (3)
Lymphocyte count decreased (Investigations) | 9 (25) | 7 (21)
Lymphocyte count increased (Investigations) | 13 (25) | 19 (35)
Neutrophil count decreased (Investigations) | 21 (117) | 24 (98)
Platelet count decreased (Investigations) | 18 (67) | 19 (66)
Weight gain (Investigations) | 2 (2) | 2 (2)
Weight loss (Investigations) | 5 (7) | 8 (13)
White blood cell decreased (Investigations) | 12 (57) | 9 (28)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (4) | 6 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 24 (94) | 24 (117)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 4 (6)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 7 (14) | 10 (37)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 6 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (22) | 9 (18)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (7) | 9 (18)
Hypokalemia (Metabolism and nutrition disorders) | 9 (27) | 10 (22)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 4 (8) | 3 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (15) | 13 (58)
Metabolism and nutrition disorders, other (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 6 (10)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 6 (7)
Musculoskeletal and connective tissue disorder, other (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 11 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (8)
Neoplasms benign, malignant and unspecified, other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (6) | 7 (9)
Dizziness (Nervous system disorders) | 5 (7) | 8 (10)
Dysesthesia (Nervous system disorders) | 7 (11) | 7 (9)
Dysgeusia (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 13 (19) | 16 (29)
Paresthesia (Nervous system disorders) | 5 (5) | 5 (5)
Presyncope (Nervous system disorders) | 1 (3) | 2 (3)
Sinus pain (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (5) | 4 (5)
Chronic kidney disease (Renal and urinary disorders) | 5 (6) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal calculi (Renal and urinary disorders) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 22 (27)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 11 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 9 (10)
Respiratory, thoracic and mediastinal disorders, other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 14 (20)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 (25) | 9 (19)
Skin and subcutaneous tissue disorders, other (Skin and subcutaneous tissue disorders) | 15 (40) | 16 (32)
Flushing (Vascular disorders) | 2 (2) | 1 (2)
Hypertension (Vascular disorders) | 23 (79) | 25 (90)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT01351896/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT01351896/ICF_001.pdf